CLINICAL TRIAL: NCT01220869
Title: An Open-label, Multi-centre Registration Trial, Investigating Efficacy and Safety of Degarelix One-month Dosing Regimen in Taiwanese Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: A Study of Degarelix in Taiwanese Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS43
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2013-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Degarelix (Experimental)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Degarelix was given as subcutaneous (s.c.) injections with a 240 mg starting dose followed one month later by a 80 mg maintenance dose. The maintenance dosing was repeated for an additional 5 months (total treatment period was 168 days).
  Other Names: degarelix acetate; Firmagon; FE200486

SUMMARY:
A phase III trial investigating the efficacy and safety of degarelix one-month depot in Taiwanese patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Has a histological confirmed prostate cancer
* Has a screening serum testosterone above 1.5 ng/mL
* Has a Eastern Cooperative Oncology Group (ECOG) score of ≤ 2
* Has a screening PSA value of ≥2 ng/mL
* Has a life expectancy of at least 168 days

Exclusion Criteria:

* Current or previous hormone therapy
* Is currently treated with 5-α-reductase inhibitor
* Has a history of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema
* Is considered to be a candidate for curative therapy, i.e radical prostatectomy or radiotherapy
* Has had cancer within the last five years except prostate cancer and surgically removed basal or squamous cell carcinoma of the skin.
* Has a clinically significant disorder (other than prostate cancer) or any other condition , including alcohol or drug abuse, which may interfere with trial participation or which may affect the conclusion of the trial as judged by the investigator
* Has received an investigational drug within the last 28 days preceding Screening Visit or longer if considered to possibly influence the outcome of the current trial

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (10):
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Medical Foundation, Chiayi Branch, Chiayi City
  - Chang Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Foundation Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkuo, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited among the patients attending the clinics included in the trial
Pre-assignment Details: 125 participants were screened and 110 participants were enrolled and exposed to degarelix.
Period: Overall Study
Arm/Group | Degarelix
Started | 110
Completed | 104
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: The number of baseline participants is identical to the number of patients exposed to degarelix.
Groups:
- Degarelix: Degarelix 240/80 mg dosing regimen (240 mg is the initiation dose, the 80 mg is the maintenance dose)
Arm/Group | Degarelix
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 110
Region of Enrollment [Number; unit: participants]
  Taiwan | 110

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of Participants With Testosterone at Castrate Level <= 0.5 ng/mL From Day 28 to Day 168
Description: Kaplan-Meier estimates of the cumulative probability of testosterone levels below castrate level (<= 0.5 ng/mL) from Day 28 to Day 168 and the associated two-sided 95% confidence interval (CI) was based on log-log transformation, Greenwood's formula, and asymptotic maximum likelihood theory. The primary objective was met if the lower limit of this two-sided 95% CI was ≥90%. The definition of the primary endpoint was the Day 28 to Day 168 cumulative probability of testosterone levels below castrate levels (≤0.5 ng/mL). Only patients with a testosterone value on Day 28 and after were included in this analysis. Patients who did not experience a testosterone suppression (≤0.5 ng/mL) were censored at the time of last available testosterone measurement. The full analysis set (FAS) results were considered primary, whereas the corresponding per protocol (PP) analysis served as the sensitivity analysis.
Time Frame: From Day 28 to Day 168
Population: The data of all participants who received at least one dose of degarelix and had at least one efficacy assessment after dosing comprised the FAS dataset.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Degarelix
Number analyzed (Participants) | 101
Percentage of participants | 97.2 [91.6 to 99.1]

2. Secondary Outcome: Proportion of Participants With Testosterone at Castrate Level (<= 0.5 ng/mL) at Day 3
Description: Proportion of participants with testosterone at castrate level (<= 0.5 ng/mL) at Day 3
Time Frame: Day 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Degarelix
Number analyzed (Participants) | 108
Percentage of participants | 93.5 [87.1 to 97.4]

3. Secondary Outcome: Percentage Change in Serum Prostate Specific Antigen (PSA) Levels From Baseline (Day 0) to Day 28
Description: Percentage change in serum prostate specific antigen (PSA levels from Baseline (Day 0) to Day 28
Time Frame: From Day 0 to Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percentage change of PSA
Arm/Group | Degarelix
Number analyzed (Participants) | 106
Percentage change of PSA | -92.4 [-96.0 to -83.6]

4. Other Pre Specified Outcome: Cumulative Probability of Participants With Testosterone at Castrate Level <= 0.5 ng/mL From Day 28 to Day 168 - Sensitivity Analysis
Description: Kaplan-Meier estimates of the cumulative probability of testosterone levels below castrate level (<= 0.5 ng/mL) from Day 28 to Day 168 and the associated two-sided 95% CI was based on log-log transformation, Greenwood's formula, and asymptotic maximum likelihood theory. The primary objective was met if the lower limit of this two-sided 95% CI was ≥90%. The definition of the primary endpoint was the Day 28 to Day 168 cumulative probability of testosterone levels below castrate levels (≤0.5 ng/mL). Only patients with a testosterone value on Day 28 and after were included in this analysis. Patients who did not experience a testosterone suppression (≤0.5 ng/mL) were censored at the time of last available testosterone measurement. The FAS analysis results were considered primary, whereas the corresponding PP analysis served as the sensitivity analysis.
Time Frame: From Day 28 to Day 168
Population: The PP analysis set included all participants from the FAS analysis set without major protocol violations.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Degarelix
Number analyzed (Participants) | 101
Percentage of participants | 97.2 [91.6 to 99.1]

5. Secondary Outcome: Cumulative Probability of no PSA Failure
Description: The time to PSA failure was defined as the days from first dosing (scheduled trial days) where an increase in serum PSA of ≥50% from nadir and at least 5 ng/mL measured on two consecutive occasions at least two weeks apart was noted. The second occasion was the time point of meeting the criterion. The Kaplan-Meier estimate and associated 95% CI were provided.
Time Frame: Day 0, Day 7, Day 28, Day 112, Day 140, Daý 168
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Degarelix
Number analyzed (Participants) | 110
Percentage of participants
  Day 0 | 100 [96.6 to 100]
  Day 0 to <= Day 7 | 100 [96.6 to 100]
  Day 0 to <= Day 28 | 100 [96.6 to 100]
  Day 0 to <= Day 112 | 99.1 [93.5 to 99.9]
  Day 0 to <= Day 140 | 98.1 [92.6 to 99.5]
  Day 0 to <= Day 168 | 96.2 [90.1 to 98.5]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signed informed consent until the end-of-trial visit, 168 days.
Description: Adverse events were evaluated at each visit.
Arm/Group | Degarelix
Serious Adverse Events (participants affected / at risk) | 9/110
Other Adverse Events (participants affected / at risk) | 69/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix (N=110)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
Oedema peripheral (General disorders) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Carcinoembryonic antigen increased (Investigations) | 1
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Bladder obstruction (Renal and urinary disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix (N=110)
Anaemia (Blood and lymphatic system disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 8 (8)
Injection site erythema (General disorders) | 31 (92)
Injection site pain (General disorders) | 27 (75)
Injection site induration (General disorders) | 18 (78)
Injection site swelling (General disorders) | 17 (20)
Hepatic function abnormal (Hepatobiliary disorders) | 10 (11)
Urinary tract infection (Infections and infestations) | 6 (7)
Dizziness (Nervous system disorders) | 7 (7)
Dysuria (Renal and urinary disorders) | 10 (10)
Hot flush (Vascular disorders) | 11 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.